CLINICAL TRIAL: NCT01109485
Title: Clinical Evaluation of 0.1% Olopatadine Hydrochloride Ophthalmic Solution in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JPN-P-2010-1
Record Dates: First submitted 2010-04-12; First posted 2010-04-23 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2011-09

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergic conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olopatadine (Experimental): Olopatadine hydrochloride ophthalmic solution 0.1%
  Interventions: Drug: Olopatadine hydrochloride ophthalmic solution 0.1%

INTERVENTIONS:
Drug: Olopatadine hydrochloride ophthalmic solution 0.1% — 1-2 drops 4 times per day

SUMMARY:
The objective of this study is to further evaluate the safety of Olopatadine Ophthalmic Solution 0.1% in Japanese children with allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose parents or guardians can issue informed consent
* Patients aged over 7 and less than 16 at the baseline
* Patients confirmed to show type I allergy
* Patients with allergic conjunctivitis
* Patients having subjective symptoms at the baseline (itching sensation, foreign body sensation, eye pain, etc.)

Exclusion Criteria:

* Patients having ocular itching sensation and injection caused by disease other than allergic conjunctivitis
* Patients having retinal detachment, diabetic retinopathy or progressive retinal disease
* Patients with a history of ocular infection, corneal herpes or relapsing corneal erosion of sudden onset or secondary to corneal injury
* Patients having received continuous treatment with corticosteroid within 3 months
* Patients having received immunotherapy
* Patients requiring continuous treatment of corticosteroid, immunosuppressors, non-steroidal anti-inflammatory agents, vasoconstrictors, anti-histamines, anti-allergy agents, herbal preparations indicated for "conjunctivitis" or any ophthalmic solution other than the test product
* Patients having undergone ocular laser therapy within 3 months
* Unilaterally blind patients (best corrected visual acuity: below 0.01)
* Patients with a history of allergy or hypersensitivity to olopatadine hydrochloride
* Patients necessitating the use of contact lens during the study period
* Other patients judged by the attending physician as inappropriate for study

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 4 weeks
Questionnaire about compliance with dosing instructions | 4 weeks
  (1;always >90% 2;often 75-90% 3;sometimes 50-75% 4;seldom <50%)

SECONDARY OUTCOMES:
Changes in score of subjective symptoms and objective findings | 4 weeks
  (0;none 1;mild 2;moderate 3;severe)
Questionnaire about stinging after instillation | 4 weeks
  (1;none 2;mild 3;moderate 4;severe)

CONTACTS AND LOCATIONS:
Overall Officials: Eriko Chono, Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center For Trial Locations, Tokyo, Japan